CLINICAL TRIAL: NCT02234440
Title: Effect of Metformin on Disease Progression in Patients With Cryptogenic Cirrhosis (NASH-related Cirrhosis) With Diabetes or Impaired Glucose Tolerance or Insulin Resistance: a Prospective Randomized, Open Labeled, Clinical Trial"
Brief Title: Effect of Metformin on Disease Progression in Patients With Cryptogenic Cirrhosis (NASH-related Cirrhosis) With Diabetes or Impaired Glucose Tolerance or Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-NASH-Cirrhosis-01
Record Dates: First submitted 2014-08-31; First posted 2014-09-09 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2016-02

CONDITIONS: NASH Related Cirrhosis
MeSH Terms: interventions — Metformin; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin- 500 mg once daily as a starting dose, can be escalated to 2 g/day to control diabetes
  Interventions: Drug: Metformin
- Insulin (Active Comparator)
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Metformin
  Arms: Metformin
Drug: Insulin
  Arms: Insulin

SUMMARY:
In this study, consecutive patients with cryptogenic cirrhosis (NASH-related cirrhosis), coming to ILBS (Institute of Liver & Biliary Sciences) OPD (Out patient Department) or getting admitted in the ward will be enrolled on fulfillment of inclusion/exclusion criteria and consent of the patient. These patients will be randomised to either metformin arm or conventional treatment arm. After enrollment these subjects will be monitored every three monthly for total of 12 months or till the primary endpoint is achieved. At the end of the study, outcome will be measured appropriately.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Patients with cryptogenic cirrhosis {NASH (Nash Alcoholic Steatohepatitis)-related cirrhosis}
3. Presence of diabetes mellitus or insulin resistance

Exclusion Criteria:

1. Patients with heart failure
2. Patients with acute kidney injury at the time of enrollment
3. Patients with CKD (Chronic Kidney Disease) or with S. Creatinine > 1 mg/dL
4. Patient with active upper GI bleeding- not settled
5. Patient with SIRS/sepsis/shock
6. Patient in ICU (Intensive Care Unit)
7. Pregnancy
8. Patients with hepatocellular carcinoma
9. Patients who are not willing to participate in the study
10. Patients with any form of decompensation at the time of enrollment in the study
11. Patient with large esophageal varices/ patients who are on beta blocker other than those patients with HVPG (Hepatic Venous Pressure Gradient) non responder to betablocker
12. Patient who has already been receiving Metformin prior to enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Reduction of portal pressure | 1 Year

SECONDARY OUTCOMES:
Improvement in fibrosis(assessed by noninvasive methods like Fibroscan and Fib 4 index) | 1 Year
Safety profile of the drugs like Random Blood Sugar (RBS) and serum lactate monitoring regularly. | 1.5 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Tanmay S Vyas, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India